CLINICAL TRIAL: NCT01952301
Title: A Randomized, Controlled Clinical Trial to Evaluate a Xenogeneic Collagen Matrix as an Alternative to Free Gingival Grafting for Oral Soft Tissue Augmentation
Brief Title: Xenogeneic Collagen Matrix as an Alternative to Free Gingival Grafting for Oral Soft Tissue Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Perio Health Professionals, PLLC (Other)
Responsible Party: Principal Investigator, Michael K McGuire, Michael K McGuire DDS, Perio Health Professionals, PLLC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13562-007
Record Dates: First submitted 2013-09-24; First posted 2013-09-27 (Estimated); Results first posted 2014-05-15 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Gingival Diseases
Keywords: Autologous; Collagen Matrix; Keratinized Tissue
MeSH Terms: conditions — Gingival Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- xenogeneic collagen matrix (Active Comparator): Xenogeneic collagen matrix device placed on treatment wound bed site
  Interventions: Device: Xenogeneic Collagen Matrix
- Free Gingival Graft (Active Comparator): Traditional free gingival graft (autogenous graft device harvested from patient's palate) placed on treatment site wound bed
  Interventions: Device: Free Gingival Graft

INTERVENTIONS:
Device: Xenogeneic Collagen Matrix — A type I and III porcine collagen matrix, as cleared by FDA (K012423)
  Arms: xenogeneic collagen matrix
Device: Free Gingival Graft — Autogenous, full-thickness soft tissue graft harvested from patient's palate.
  Other Names: Free Autogenous Graft
  Arms: Free Gingival Graft

SUMMARY:
A split-mouth study comparing soft tissue augmentation results using free gingival graft (FGG) versus xenogeneic collagen matrix (CM) for the generation of keratinized tissue (KT) around teeth with insufficient (< 2mm) KT.

DETAILED DESCRIPTION:
A single-blind, randomized, controlled, split-mouth study of 30 subjects with insufficient zones of KT (< 2mm). The study utilized a within subject treatment comparison design to establish non-inferiority of the test (CM) versus control (FGG) therapy. The primary efficacy endpoint was KT width at 6-months. Secondary endpoints included traditional periodontal measures, such as clinical attachment, recession and bleeding on probing. Patient reported pain, discomfort and esthetic satisfaction were also recorded. Biopsies were obtained at 6-months.

ELIGIBILITY:
Inclusion Criteria:

* At least two non-adjacent teeth in contralateral quadrants of the same jaw with < 2mm of KT that requires soft tissue grafting (1-4 teeth may be treated). In case of adjacent teeth requiring grafting, only one tooth at each site will act as test or control tooth, but all teeth will get the same treatment). The number of teeth treated must be the same on the test and control sites.

  * Root coverage is not desired at the time of grafting.
  * Females of childbearing potential must have a documented negative urine pregnancy test.
  * Read, understood and signed an institutional review board (IRB) approved Informed Consent Form (ICF).
  * Able and willing to follow study procedures and instructions.
  * Multi-rooted teeth may be treated but will not be included as study teeth

Exclusion Criteria:

* Vestibule depth of less than 7mm from base of recession, and/or teeth with Miller Grade 2 or higher mobility.

  * Any systemic conditions (i.e., diabetes mellitus, cancer, HIV, bone metabolic diseases) that could compromise wound healing and/ or preclude periodontal surgery; or who are currently receiving or have received within two months prior to study entry, systemic corticosteroids, immunosuppressive agents, radiation therapy, and/or chemotherapy which could compromise wound healing and preclude periodontal surgery.
  * Presence of acute infectious lesions in the areas intended for surgery.
  * History of any tobacco use within the last six months.
  * Taking intramuscular or intravenous bisphosphonates.
  * Known hypersensitivity to collagen products, and/or allergy to iodine or shellfish.
  * Participating in other clinical studies involving therapeutic intervention (either medical or dental).
  * Previously undergone a gingival grafting procedure on the test or control teeth or the teeth adjacent to the study site.
  * Female subjects who are pregnant or lactating, or who intend to become pregnant during the study duration following entrance into the study.
  * Subjects, who in the opinion of the investigator, for any reason other than those listed above, will not be able to complete the study per protocol.

Ages: 8 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael K McGuire, DDS, Principal Investigator — Perio Health Professionals

REFERENCES:
- [Derived] McGuire MK, Scheyer ET. Randomized, controlled clinical trial to evaluate a xenogeneic collagen matrix as an alternative to free gingival grafting for oral soft tissue augmentation. J Periodontol. 2014 Oct;85(10):1333-41. doi: 10.1902/jop.2014.130692. Epub 2014 Mar 5. PMID 24597764

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Our study sample was derived from the population of patients who presented at our practice between 11-3-2010 and 3-16-2011 and met predetermined selection criteria
Groups:
- XCM Versus FGG: xenogeneic collagen matrix versus free gingival graft
Period: Overall Study
Arm/Group | XCM Versus FGG
Started | 30 (We designed and implemented a single-blind, randomized, controlled, split-mouth study of 30 subjects)
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Xenogeneic Collagen Matrix Versus Free Gingival Graft: free gingival graft versus a xenogeneic collagen matrix over an apically positioned flap used to generate keratinized tissue
Arm/Group | Xenogeneic Collagen Matrix Versus Free Gingival Graft
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Keratinized Tissue Width
Description: Change in Keratinized Tissue width
Time Frame: 6 months
Population: Sample size was determined using 80% power fans assuming a paired t-test of non-inferiority with a non-inferiority margin of 1.0 mm, a within-subject standard deviation of 1.0 mm, and a one-sided alpha of 0.05, resulting in a sample size of 27. To account for potential loss-to-follow-up, 30 subjects were enrolled in the trial.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Free Gingival Graft: free gingival graft over an apically positioned flap used to generate keratinized tissue
- Xenogeneic Collagen Matrix: xenogeneic collagen matrix over an apically positioned flap to generate keratinized tissue
Arm/Group | Free Gingival Graft | Xenogeneic Collagen Matrix
Number analyzed (Participants) | 30 | 30
mm | 4.42 (0.64) | 2.92 (0.88)
Statistical Analysis 1: Comparison: Free Gingival Graft vs Xenogeneic Collagen Matrix; Test type: Non-Inferiority or Equivalence — The primary hypothesis of the study evaluated whether CM was not inferior to Control in the generation of KT width from baseline to 6 months. A paired t-test was used to test for non-inferiority, using a one-sided significance level of 0.05 and a non-inferiority margin of 1.0 mm; p < 0.0001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Xenogeneic Collagen Matrix: xenogeneic collagen matrix over an apically positioned flap used to generate keratinized tissue
Arm/Group | Free Gingival Graft | Xenogeneic Collagen Matrix
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No